CLINICAL TRIAL: NCT01309074
Title: Does Pregabalin Improve Symptoms of Anxiety in Patients With Epilepsy? A Comparison With Sertraline
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No subjects could be enrolled and therefore we decided to withdraw/stop the study.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GA0082BY
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy; Anxiety
Keywords: Anxiety; Epilepsy
MeSH Terms: conditions — Epilepsy; Anxiety Disorders | interventions — Pregabalin; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin is an antiepileptic medication which has been found in double blind placebo controlled trials to be effective and safe in the treatment of primary generalized anxiety disorder. It has an indication for the treatment of this condition in Europe & Canada but not in the US.
  Interventions: Drug: Pregabalin-Lyrica
- Sertraline (Active Comparator): Sertraline is an SSRI found to be an effective treatment of generalized anxiety disorder in controlled trials. It does not have an indication for this in this country.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Pregabalin-Lyrica — Pregabalin in a dose up to 300mg/day in BID dosing.
  Other Names: Lyrica.
  Arms: Pregabalin
Drug: Sertraline — Sertraline in a dose up to 200mg/day in BID dosing.
  Other Names: Zoloft.
  Arms: Sertraline

SUMMARY:
The aim of the study is to compare the safety & efficacy of sertraline (up to a dose of 200mg/day) & pregabalin (up to a dose of 300mg/day) for the treatment of symptoms of anxiety in patients with epilepsy.

DETAILED DESCRIPTION:
Patients with epilepsy will be treated with either sertraline (up to a dose of 200mg/day) or pregabalin (up to a dose of 300mg/day) for the treatment of symptoms of anxiety. Outcome measures will include changes in the anxiety severity scales.

ELIGIBILITY:
Inclusion Criteria:

* GAD-7 total score above 10.
* Have a diagnosis of a Partial Seizure Disorder.
* Have a Hamilton-A total score 20 and above.
* 18-80 years of age.
* Able to read at a fourth grade level.
* If a woman of childbearing age, agrees to use an acceptable means of birth control.

Exclusion Criteria:

* Unable to understand and sign a consent.
* Unable to follow instructions for the study.
* Displaying current suicidal ideation
* Having psychogenic non-epileptic seizures
* Have a history of drug or alcohol abuse.
* Use of any investigational drug within the last 30 days.
* Hypersensitivity reaction or other serious adverse event to PGB in prior trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement of anxiety symptoms measured with the changes of the total scores of GAD-7 & HAM-A. | 27 weeks
  Change in severity of symptoms &/o remission of symptoms of anxiety between visit 0 & the end of treatment phase.

SECONDARY OUTCOMES:
Change in Quality of life measures assessed with the QOLIE-89. | 27 weeks.
  A change in the total scores of the QOLIE-89 scores as well as in the individual subscales and change in the tolerance of antiepileptic medication assessed with change in the total score of the adverse event profile between baseline & the end of treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Andre M. Kanner, MD, Principal Investigator — Director Laboratory Encephalography
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States